CLINICAL TRIAL: NCT06147674
Title: Evaluation of VQm Pulmonary Health Monitor™ on Pulmonary Health Parameters for Intensive Care Medicine
Brief Title: Evaluation of VQm PHM on Pulmonary Health Parameters for ICU
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Rostrum Medical Innovations Inc. (Industry)
Collaborators: Medical Initiatives (Network)
Responsible Party: Sponsor
Other Study IDs: LM02-CLR-0002
Record Dates: First submitted 2023-07-26; First posted 2023-11-27 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Ventilators, Mechanical; Stroke; COPD; Acute Lung Injury/Acute Respiratory Distress Syndrome (ARDS); Pneumonia
Keywords: Ventilation; ICU; Cardiopulmonary health
MeSH Terms: conditions — Stroke; Pulmonary Disease, Chronic Obstructive; Acute Lung Injury; Respiratory Distress Syndrome; Pneumonia; Respiratory Aspiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- VQm PHM™: Non-invasive measurements obtained with the VQm PHM™ compared to current standard of care.
  Interventions: Device: VQm Pulmonary Health Monitor™

INTERVENTIONS:
Device: VQm Pulmonary Health Monitor™ — The VQm Pulmonary Health Monitor™ (may be referred to as the VQm PHM™) is a a Class IIa, Health Canada approved medical device used as an adjunct monitor and is non-life supporting, providing clinicians with measurements of pulmonary function parameters of mechanically ventilated adult patients. The measurements provided are:
  * Pulmonary Blood Flow (PBF)
  * Shunt Fraction (Qsi)
  * Dead space (VD):
  * Functional Residual Capacity (FRC)

SUMMARY:
The goal of this observational study is to compare pulmonary health parameter measurements from the VQm PHM™ to existing clinical measurements. The main questions it aims to answer are:

* Confirm the performance of non-invasive pulmonary health parameter shunt fraction value found on the VQm PHM™ when compared to available reference measurements.
* Confirm the performance of non-invasive pulmonary health parameter pulmonary blood flow, functional residual capacity and physiological dead space found on the VQm PHM™ when compared to available reference measurements.

DETAILED DESCRIPTION:
This is a multi-site, international, prospective, non-blinded, non-randomized, observational study. This study aims to compare measurements from the VQm PHM™ to existing clinical measurements, assess safety of the device and determine effects that standard clinical events have on the VQm PHM™ measurements. This study does not include changes to clinical care based on measurements from the VQm PHM™. Each patient will serve as their own control.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 years old or above, at the time of the inclusion
* Patient currently admitted in the ICU, who are indicated for cardiac output monitoring using a pulmonary artery catheter and who require pressure or volume controlled mechanical ventilation using an ETT
* Provision of signed and dated informed consent form (ICF) by the patient or a trusted person

Exclusion Criteria:

* Male or female under the age of 18 years old, at the time of screening
* Patient under guardianship
* Patient who requires tidal volumes of less than 250cc
* Pregnancy
* Patient whose care requires the use of an anesthetic conserving device
* Patient whose care requires a closed-loop ventilator
* Patient who is unable to tolerate a transient increase in inhaled CO2
* Patient who is unable to tolerate a transient inhalation of N2O or is contraindicated to N2O use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients currently admitted to the ICUs requiring mechanical ventilation will be screened for potential enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-01-15 (Estimated); Primary Completion 2025-01-15 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Shunt fraction value | Through study completion, an average of 12 months
  Confirming the performance of non-invasive pulmonary health parameter shunt value found on the VQm PHM™ monitor when compared to available reference measurements

SECONDARY OUTCOMES:
Pulmonary blood flow - trend | Through study completion, an average of 12 months
  Confirming the performance of non-invasive pulmonary health parameter PBF trend found on the VQm PHM™ monitor when compared to available reference measurements
Functional residual capacity - trend | Through study completion, an average of 12 months
  Confirming the performance of non-invasive pulmonary health parameter FRC trend found on the VQm PHM™ monitor when compared to available reference measurements
Pulmonary blood flow - absolute value | Through study completion, an average of 12 months
  Confirming the performance of non-invasive pulmonary health parameter PBF absolute values found on the VQm PHM™ monitor when compared to available reference measurements
Functional residual capacity - absolute value | Through study completion, an average of 12 months
  Confirming the performance of non-invasive pulmonary health parameter FRC absolute values found on the VQm PHM™ monitor when compared to available reference measurements
Physiological dead space | Through study completion, an average of 12 months
  Confirming the performance of non-invasive pulmonary health parameter physiological dead space value found on the VQm PHM™ monitor when compared to available reference measurements
Oxygen desaturation due to breathing circuit connectivity (safety) | Through completion of study, up to 72 horus
  Number of participants with treatment-related adverse events due to faulty connecting the breathing circuit during normal operation the VQm PHM™ monitor as measured by oxygen saturation desaturations of SpO2 <89% for >14s.
High pressure due to volume control (safety) | Through completion of study, up to 72 hours
  Number of participants with device-related adverse events due to increased pressure induced by volume-control mode as determined by peak pressure >10cm H2O ventilator setting.
High volume due to pressure control (safety) | Through completion of study, up to 72 hours
  Number of participants with device-related adverse events due to increased volume induced by pressure-control mode as determined by a volume >200mL from target volume.
Safe range of nitrous oxide delivery (safety) | Through completion of study, up to 72 hours
  Confirming the acceptable safety limitations of nitrous oxide gas delivery by the VQm PHM™ monitor below 10% as measured by the device.
Incident rate of adverse events, adverse events and treatment-emergent serious adverse events | Through completion of study, up to 72 hours
  As deemed caused by the the VQm PHM™ monitor during standard of care in the ICU setting.

OTHER OUTCOMES:
Shunt fraction changes due to ETT Clamping | Through completion of study, up to 72 hours
  Determining the effects of clamping the ETT on shunt fraction compared to baseline
PBF changes due to ETT Clamping | Through completion of study, up to 72 hours
  Determining the effects of clamping the ETT on PBF compared to baseline
FRC changes due to ETT Clamping | Through completion of study, up to 72 hours
  Determining the effects of clamping the ETT on FRC compared to baseline
VD changes due to ETT Clamping | Through completion of study, up to 72 hours
  Determining the effects of clamping the ETT on VD compared to baseline
Shunt fraction changes due to participant positional changes | Through completion of study, up to 72 hours
  Determining the effects of positional changes [i.e. passive leg raise, semi-recumbent] the pulmonary health parameters (shunt fraction) compared to baseline
PBF changes due to participant positional changes | Through completion of study, up to 72 hours
  Determining the effects of positional changes [i.e. passive leg raise, semi-recumbent] the pulmonary health parameters (PBF) compared to baseline
FRC changes due to participant positional changes | Through completion of study, up to 72 hours
  Determining the effects of positional changes [i.e. passive leg raise, semi-recumbent] the pulmonary health parameters (FRC) compared to baseline
VD changes due to participant positional changes | Through completion of study, up to 72 hours
  Determining the effects of positional changes [i.e. passive leg raise, semi-recumbent] the pulmonary health parameters (VD) compared to baseline
Shunt fraction changes due to delivery of vasopressors | Through completion of study, up to 72 hours
  Determining the effects of vasopressor administration on the pulmonary health parameters (shunt fraction) compared to baseline
PBF changes due to delivery of vasopressors | Through completion of study, up to 72 hours
  Determining the effects of vasopressor administration on the pulmonary health parameters (PBF) compared to baseline
FRC changes due to delivery of vasopressors | Through completion of study, up to 72 hours
  Determining the effects of vasopressor administration on the pulmonary health parameters (FRC) compared to baseline
VD changes due to delivery of vasopressors | Through completion of study, up to 72 hours
  Determining the effects of vasopressor administration on the pulmonary health parameters (VD) compared to baseline
Shunt fraction changes due to progression of ARDS | Through completion of study, up to 72 hours
  Determining the effects of ARDS on the pulmonary health parameters (shunt fraction) compared to baseline
PBF changes due to progression of ARDS | Through completion of study, up to 72 hours
  Determining the effects of ARDS on the pulmonary health parameters (PBF) compared to baseline
FRC changes due to progression of ARDS | Through completion of study, up to 72 hours
  Determining the effects of ARDS on the pulmonary health parameters (FRC) compared to baseline
VD changes due to progression of ARDS | Through completion of study, up to 72 hours
  Determining the effects of ARDS on the pulmonary health parameters (VD) compared to baseline

CONTACTS AND LOCATIONS:
Locations (4):
- UC Davis Medical Center, Sacramento, California, United States
- Medical University of Vienna, Vienna, Austria
- University Hospital Kralovske Vinohrady, Prague, Czechia
- Hôpital Européen Georges Pompidou, Paris, France

IPD SHARING:
Plan to Share IPD: No